CLINICAL TRIAL: NCT00488722
Title: A Prospective, Single-Arm Study to Evaluate the Efficacy and Safety of Zoladex 3.6mg Combined With CEF Chemotherapy as Neo-Adjuvant Therapy in Hormone Responsive, Premenopausal, Operable Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: jzhang
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer
Keywords: To observe the biological changes under concurrent Zoladex and CEF as neoadjuvant regimen with respect to the ER,PR,cerbB-2 status before and after therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zoladex

SUMMARY:
It has been found that many breast cancers are hormone dependent and that hormonal therapy by estrogen suppression such as ovarian ablation, tamoxifen and aromatase inhibitor has proven beneficial in both adjuvant and neoadjuvant settings. Zoladex, a kind of luitinizing hormone releasing hormone analogue, can offer efficient estrogen suppression as well. It can induce reversible amenorrhea and the clinical effect is similar to ovarian ablation. Some studies have demonstrated the efficacy of zoladex in treating pre and perimenopausal hormone dependent breast cancer in both adjuvant and metastatic settings. Few data is available on Zoladex in neoadjuvant treatment for breast cancer In our departments, neoadjuvant CEF regimen is of general practice, and a preliminary study is designed to investigate whether adding Zoladex into neoadjuvant CEF could further improve results in hormone responsive breast cancer.

DETAILED DESCRIPTION:
It has been found that many breast cancers are hormone dependent and that hormonal therapy by estrogen suppression such as ovarian ablation, tamoxifen and aromatase inhibitor has proven beneficial in both adjuvant and neoadjuvant settings. Zoladex, a kind of luitinizing hormone releasing hormone analogue, can offer efficient estrogen suppression as well. It can induce reversible amenorrhea and the clinical effect is similar to ovarian ablation. Some studies have demonstrated the efficacy of zoladex in treating pre and perimenopausal hormone dependent breast cancer in both adjuvant and metastatic settings. Few data is available on Zoladex in neoadjuvant treatment for breast cancer In our departments, neoadjuvant CEF regimen is of general practice, and a preliminary study is designed to investigate whether adding Zoladex into neoadjuvant CEF could further improve results in hormone responsive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Pathological confirmation of breast cancer
3. Tumor stage(TNM):T2-4bN0-3M0
4. ER(+) and/or PR(+).
5. Premenopausal woman.
6. Age≥40 years
7. Measurable disease as per RECIST criteria
8. Karnofsky≥70
9. Labratory criteria:

   * PLT≥100*109/L
   * WBC≥4000/mm3
   * HGB≥10g/dl
   * ALT and AST<2*ULN

Exclusion Criteria:

1. Presence of metastatic disease.
2. Inflammatory breast cancer.
3. Bilateral breast cancer.
4. previous chemotherapy or hormonal therapyfor current breast neoplasm.
5. other malignant tumor (concurrent or previous).
6. Pregnant woman.
7. Hypersensitive to any drug in CEF regimen or any ingredient of Zoladex.
8. Any severe systemic disease contraindicating chemotherapy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-04; Study Completion 2009-03

PRIMARY OUTCOMES:
To evaluate the efficacy of concurrent Zoladex and CEF as neoadjuvant regimen in terms of: ORR(CR+PR) and PCR

SECONDARY OUTCOMES:
To evaluate the efficacy of concurrent Zoladex and CEF as neoadjuvant regimen in terms of: CBR, downstaging rates in tumor size and axillary lymph node -To evaluate the safety of concurrent Zoladex and CEF as neoadjuvant regimen

CONTACTS AND LOCATIONS:
Overall Officials: ZHNAG JIN, PROFESSOR, Principal Investigator — Tianjin Cancer Hospital; ZHANG JIN, PROFESSOR, Principal Investigator — TAINJIN CANCER HOSPITAL
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhang S, Zhang C, Liu J, Qin L, Cui S, Zhang J. A Phase II trial of Zoladex combined with CEF chemotherapy as neoadjuvant therapy in premenopausal women with hormone-responsive, operable breast cancer. Med Oncol. 2012 Jun;29(2):479-85. doi: 10.1007/s12032-011-9883-2. Epub 2011 Mar 6. PMID 21380781